CLINICAL TRIAL: NCT06964776
Title: A Phase 1 Study to Further Investigate the Pharmacokinetics, Safety and Tolerability, Food Effect and Drug-Drug Interaction of LY4268989 (MORF-057) in Healthy Participants
Brief Title: A Study of LY4268989 (MORF-057) in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27387; J6E-MC-KWAC (Other: Eli Lilly and Company); MORF-057 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 1, 4 and 5 are blinded while Cohort 2, 3, 6, 7, and 8 are open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- LY4268989 or Placebo Cohort 1 (Blinded) (Experimental): Participants will receive LY4268989 orally or placebo single dose followed by BID administration
  Interventions: Drug: LY4268989; Drug: Placebo
- LY4268989 Cohort 2 (Open-Label) (Experimental): Participants will receive LY4268989 orally tablet (formulation compared to capsule formulation) in a fasted state
  Interventions: Drug: LY4268989
- LY4268989 Cohort 3 (Open-Label) (Experimental): Participants will receive multiple doses of LY4268989 orally BID administration with midazolam orally and intravenously (IV).
  Interventions: Drug: LY4268989; Drug: Midazolam
- LY4268989 or Placebo Cohort 4 (Blinded) (Experimental): Participants will receive single escalating doses of LY4268989 orally or placebo
  Interventions: Drug: LY4268989; Drug: Placebo
- LY4268989 Cohort 5 (Blinded) (Experimental): Participants will receive multiple doses of LY4268989 orally or placebo
  Interventions: Drug: LY4268989; Drug: Placebo
- LY4268989 Cohort 6 (Open-Label) (Experimental): Participants will receive LY4268989 single dose orally in a fasted and fed state
  Interventions: Drug: LY4268989
- LY4268989 Cohort 7 (Open-Label) (Experimental): Participants will receive multiple doses of LY4268989 orally BID administration in a fed state
  Interventions: Drug: LY4268989
- LY4268989 Cohort 8 (Open-Label) (Experimental): Participants will receive multiple doses of LY4268989 orally BID administration with midazolam IV in a fasted state.
  Interventions: Drug: LY4268989; Drug: Midazolam

INTERVENTIONS:
Drug: LY4268989 — Administered orally
Drug: Placebo — Administered placebo
  Arms: LY4268989 Cohort 5 (Blinded); LY4268989 or Placebo Cohort 1 (Blinded); LY4268989 or Placebo Cohort 4 (Blinded)
Drug: Midazolam — Administered orally
  Arms: LY4268989 Cohort 3 (Open-Label)
Drug: Midazolam — Administered intravenously (IV)
  Arms: LY4268989 Cohort 3 (Open-Label); LY4268989 Cohort 8 (Open-Label)

SUMMARY:
The purpose of this study is to measure the body's absorption and processing of the study drug, the study drug's effect on the body, safety, and tolerability with LY4268989 (MORF-57) in healthy participants, including Japanese and Chinese participants

ELIGIBILITY:
Inclusion Criteria:

* Are healthy as determined by medical evaluation including medical history, physical examination, laboratory test, electrocardiograms (ECGs), and vital signs.
* Cohort 5 includes Japanese participants. To qualify, the participants must be first-generation Japanese in the US, defined as the participant's biological parents, and all the participant's biological grandparents, being of exclusive Japanese descent, and being born in Japan.
* Cohort 5 includes Chinese participants. To qualify as Chinese for this study, all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China.
* Have a body mass index within the range of 18.0 to 32.0 kilogram/square meter (kg/m²), inclusive, at screening.

Exclusion Criteria:

* Have a current or recent acute, active infection. For at least 30 days before screening and up to Day 1, participants must have no symptoms or signs of confirmed or suspected infection, and must have completed any appropriate anti-infective treatment.
* Have presence of significant uncontrolled respiratory, cerebrocardiovascular, cardiovascular, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic or psychiatric disorders, or abnormal laboratory values at screening that, in the opinion of the sponsor or investigator, pose an unacceptable risk to the participant if participating in the study or of interfering with the interpretation of data.
* Are immunocompromised to an extent that participation in the study would pose an unacceptable risk to the participant as determined by the investigator.
* Use or intend to use prescription or nonprescription medication, including dietary supplements, vitamins, herbal supplements, traditional Chinese medicine, or alternative medicines, within 14 days or 5 half-lives (whichever is longer), prior to dosing, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4268989 (Cohort 1) and (Cohort 5) | Day 1 to Day 17
PK: Area Under the Concentration Curve (AUC) of LY4268989 (Cohort 1) and (Cohort 5) | Day 1 to Day 17
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) (Cohort 1), (Cohort 3), and (Cohort 5) | Baseline to Study Completion (Up to Day 17)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module
Number of Participants with TEAEs and SAEs (Cohort 4) | Baseline to Study Completion (Up to Period 4, Day 4)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the reported adverse events module
PK: Cmax of LY4268989 (Cohort 2) | Day 1 to Day 13
PK: AUC of LY4268989 (Cohort 2) | Day 1 to Day 13
PK: AUC of Midazolam and 1'-Hydroxymidazolam (Cohort 3) | Day 1 to Day 17
  PK of midazolam and 1'-hydroxymidazolam (AUC), where midazolam is administered alone and in the presence of LY4268989
PK: AUC of Midazolam and 1'-Hydroxymidazolam (Cohort 8) | Day 3 and Day 11
  PK of midazolam and 1'-hydroxymidazolam (AUC), where midazolam is administered alone and in the presence of LY4268989
PK: Cmax of Midazolam and 1'-Hydroxymidazolam (Cohort 3) | Day 1 to Day 17
  PK of midazolam and 1'-hydroxymidazolam (Cmax), when midazolam is administered alone and in the presence of LY4268989
PK: Cmax of Midazolam and 1'-Hydroxymidazolam (Cohort 8) | Day 3 to Day 11
  PK of midazolam and 1'-hydroxymidazolam (Cmax), when midazolam is administered alone and in the presence of LY4268989
PK: Cmax of LY4268989 (Cohort 6) | Day 1 to Day 7
PK: AUC of LY4268989 (Cohort 6) | Day 1 to Day 7
PK: Cmax of LY4268989 (Cohort 7) | Day 1 to Day 12
PK: AUC of LY4268989 (Cohort 7) | Day 1 to Day 12

SECONDARY OUTCOMES:
PK: Cmax of LY4268989 (Cohort 4) | Day 1 to Day 4
PK: AUC of LY4268989 (Cohort 4) | Day 1 to Day 4
PK: Cmax of LY4268989 (Cohort 3) | Time Frame: Day 6 to Day 15
PK: AUC of LY4268989 (Cohort 3) | Time Frame: Day 6 to Day 15
PK: Cmax of LY4268989 (Cohort 8) | Time Frame: Day 3 and Day 10
PK: AUC of LY4268989 (Cohort 8) | Time Frame: Day 3 and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- CenExel ACT, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No